CLINICAL TRIAL: NCT00207805
Title: The Optimal Timing of a Second Autologous Peripheral Blood Stem Cell Transplantation in Patients (<61 Years) With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre National de Greffe de Moelle Osseuse (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Procedure: autologous PBSC transplant — optimal timining of a second autologous transplant

SUMMARY:
Autologous peripheral blood stem cell (PBSC) transplantation is now considered standard therapy in patients (< 65 ans) with multiple myeloma. The Intergroupe Francophone du Myelome conducted a randomised trial of the treatment of multiple myeloma with high dose chemotherapy followed by either one or two successive autologous stem cell transplantation. The probabilities of event-free-survival and overall survival were doubled with a double transplant. The benefits were greatest among patients who had not had a very good partial response to the first transplant.

The aim of this multicenter randomised trial in previously untreated patients with multiple myelome (stage II, III DS)is to assess the optimal timing of a second autologous stem-cell transplant.After a first-line therapy with thalidomide-dexamethasone followed by a PBSC collection, patients are randomly assigned to receive two autologous PBSC transplants (arm A)or one autologous PBSC transplant followed by a consolidation therapy with thalidomide-dexamethasone (arm B). Patients included in the arm B will receive a second transplant in case of disease progression on consolidation therapy, or in case of relapse in responders.

ELIGIBILITY:
Inclusion Criteria:

* patients less than 61 years of age
* Durie Salmon stage II or III
* written and informed consent

Exclusion Criteria:

* Prior treatment for myeloma
* ECOG performance score of 4
* Positive HIV test
* Chronic respiratory disease (DLco < 60%)
* Systolic ejection fraction < 50%
* Pregnant or nursing women

Max Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202
Dates: Start 2003-05

PRIMARY OUTCOMES:
Overall survival (from randomistion) of the 2 groups at 5 years

SECONDARY OUTCOMES:
Event-free-survival

CONTACTS AND LOCATIONS:
Overall Officials: abderrahman abdelkefi, Principal Investigator — Centre National de Greffe de Moelle Osseuse; abderrahman abdelkefi, MD, Principal Investigator — Centre National de Greffe de Moelle Osseuse
Locations (1):
- Centre National de Greffe de Moelle Osseuse, Tunis, Tunisia

REFERENCES:
- [Result] Abdelkefi A, Torjman L, Ben Romdhane N, Ladeb S, El Omri H, Ben Othman T, Elloumi M, Bellaj H, Lakhal A, Jeddi R, Aissaoui L, Saad A, Hsairi M, Boukef K, Dellagi K, Ben Abdeladhim A. First-line thalidomide-dexamethasone therapy in preparation for autologous stem cell transplantation in young patients (<61 years) with symptomatic multiple myeloma. Bone Marrow Transplant. 2005 Aug;36(3):193-8. doi: 10.1038/sj.bmt.1705050. PMID 15968290 (Retraction: PMID 19513083 Bone Marrow Transplant. 2009 Jun;43(11):893)
- [Derived] Abdelkefi A, Ladeb S, Torjman L, Othman TB, Lakhal A, Romdhane NB, Omri HE, Elloumi M, Belaaj H, Jeddi R, Aissaoui L, Ksouri H, Hassen AB, Msadek F, Saad A, Hsairi M, Boukef K, Amouri A, Louzir H, Dellagi K, Abdeladhim AB; Tunisian Multiple Myeloma Study Group. Single autologous stem-cell transplantation followed by maintenance therapy with thalidomide is superior to double autologous transplantation in multiple myeloma: results of a multicenter randomized clinical trial. Blood. 2008 Feb 15;111(4):1805-10. doi: 10.1182/blood-2007-07-101212. Epub 2007 Sep 17. PMID 17875806 (Retraction: PMID 19520824 Abdelkefi A, Ladeb S, Torjman L, Ben Othman T, Lakhal A, Ben Romdhane N, Elloumi M, Jeddi R, Aissaouï L, Ben Hassen A, Msadek F, Saad A, Hsaïri M. Blood. 2009 Jun 11;113(24):6265)